CLINICAL TRIAL: NCT03613012
Title: Pain Index Extracted From EEG in Monitoring Chronic Pain
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, yifeng, Chief Physician, Peking University People's Hospital
Other Study IDs: RMYYMZK-5590
Record Dates: First submitted 2018-07-11; First posted 2018-08-02 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Chronic Pain; Pain Assessment
Keywords: Pain assessment; electroencephalographic; numerical rating scale; pain index
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pain index: Pain index will be extracted from the EEG of chronic pain patients before and after pain treatments
  Interventions: Diagnostic Test: Pain index

INTERVENTIONS:
Diagnostic Test: Pain index — Record the patients' EEG and extract pain index before and after pain treatments

SUMMARY:
Pain is a subjective feeling,and pain experts have been trying to assess it using objective methods. Pain index (PI) is extracted from electroencephalographic as an objective diagnostic tool for chronic pain. This study is a diagnostic test aims to explore the reliability and validity of PI, with numerical rating scale(NRS) as the gold standard.

DETAILED DESCRIPTION:
Chronic pain outpatients between 18 and 80 years old, NRS ≥4 at first visit and receive injection or shockwave therapy will be included. After informed consents signed, the age, gender, dominant hand and hospital anxiety and depression scale (HADS) will be collected. Each patient will be connected with a multifunctional monitor HXD-1 for 8 minutes to access EEG in a quiet environment before pain treatment and 30 minutes after pain treatment. NRS will also be recorded before pain treatment and 30 minutes after pain treatment. PI will be extracted from EEG by analysts.

In order to reduce environmental effects, the same quiet research environment will be used throughout the study. All data will be obtained and recorded by the same person, and all PI will be analyzed and calculated by the same person.

SPSS 20.0 will be used to analyze the data, Pearson's correlations and Kappa consistency test to analyze the validity and reliability of PI. The receiver operating characteristic curve will be use to analyze the sensitivity and specificity of PI to evaluating moderate and severe pain(NRS≥4). A multiple linear regression equation with PI as dependent variable and anxiety score and depression score as independent variables will be used to evaluate the influence of anxiety and depression on PI.

ELIGIBILITY:
Inclusion Criteria:

* 1.chronic pain patients diagnosed lumbar disc herniation, osteoarthritis or other chronic pain diseases, who will received injection therapy or shockwave therapy at clinic.
* 2.patients age 18-80 years-old
* 3.patients with an NRS pain score ≥ 4,
* 4.patients who voluntarily participate in the test and sign the informed consent forms.

Exclusion Criteria:

* 1.patients with central nervous system disorders, such as epilepsy, cerebral infarction, or cerebral hemorrhage,
* 2.patients with mental disorders,
* 3.patients with a history of long-term use of psychotropic drugs.
* 4.patients who can't understand NRS.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample capacity calculation is based on the sensitivity/specificity of the diagnostic test allowed a minimum sensitivity of 80%, a minimum specificity of 80%, a significance level α of 0.01, an allowable error of 0.1 strictly.The estimated sample is 107 patients. Considering a predicted shedding rate of 10%, 118 patients will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Pain index | 30 mins after treatment
  Pain index is extracted from EEG accessed by a multifunctional monitor HXD-1

SECONDARY OUTCOMES:
Hamilton Anxiety and Depression Scale(HADS) | baseline
  Validated Chinese version of Hamilton Anxiety and Depression Scale is completed by the trained doctor.The HAD scale contains two sub-scales of anxiety and depression, consisting of 14 items, of which 7 items are rated as depression, 7 items are assessed as anxiety.Each item is scored from 0 to 3 points.Therefore, the anxiety subscale ranges from 0 to 21,and higher values represent a worse outcome: 0~7:asymptomatic, 8~10:suspicious presence; 11 to 21: existed.The depression subscale is scored in the same way as the anxiety scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No